CLINICAL TRIAL: NCT03663231
Title: Duration of Effect of Biotene Spray in Patients With Symptomatic Dry Mouth
Brief Title: Duration of Effect of Biotene Spray in Patients With Dry Mouth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Ralph Saunders, Professor, University of Rochester
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69726
Record Dates: First submitted 2018-08-08; First posted 2018-09-10 (Actual); Results first posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-12

CONDITIONS: Dry Mouth
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Biotene (Experimental): People who present with dry mouth and will receive a single dose of Biotene.
  Interventions: Device: Biotene
- Placebo (Placebo Comparator): People who present with dry mouth and will receive a single dose of an alternative agent.
  Interventions: Device: Placebo

INTERVENTIONS:
Device: Biotene — Biotène Dry Mouth Moisturizing Spray contains water, polyglycitol, propylene glycol, sunflower oil, xylitol, milk protein extract, potassium sorbate, acesulfame K, potassium thiocyanate, lysozyme, lactoferrin, lactoperoxidase. 3 sprays, approximately 15 mL.
  Arms: Biotene
Device: Placebo — IND/IDE exempt device primarily water
  Arms: Placebo

SUMMARY:
To determine the duration of effect of a single dose of Biotène Moisturizing Mouth Spray in subjects who complain of a clinically dry mouth. The effect of the product will be compared to a control spray (water).

ELIGIBILITY:
Inclusion Criteria:

* Adults who are in good general health and reply initially affirmatively to the question, "Do you feel that your mouth is too dry and causes you discomfort at times during the day other than on awakening from sleep?" This question is an adaptation of the question used successfully by Jose and others (2016) to recruit study subjects.
* Adults who are able to communicate easily in English and who are able to demonstrate understanding of the study instructions.
* Adults who are physically able to perform an unstimulated whole saliva flow rate (UWSFR) test and who produce 0.2 mL/min or less of saliva.

Exclusion Criteria:

* Adults under the care of a health professional specifically for xerostomia treatment, including those taking prescription systemic parasympathetic medications.
* Adults who regularly "self-medicate" their xerostomia with water or other agents or products designed to treat their xerostomia and are unwilling or unable to cease use of the agent for at least 48 hours prior to the two test visits.
* Adults who are primarily mouth breathers (i.e. mouth breathing secondary to nasal obstruction)
* Adults who cannot consent for themselves or have physical/mental disabilities requiring a caregiver.
* Adults with a known allergy to any of the ingredients in Biotène Spray (eg. dairy allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2019-02-11 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Eastman Dental Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lung CB, Watson GE, Verma S, Feng C, Saunders RH. Duration of effect of Biotene spray in patients with symptomatic dry mouth: A pilot study. Oral Surg Oral Med Oral Pathol Oral Radiol. 2021 Apr;131(4):415-421. doi: 10.1016/j.oooo.2020.12.002. Epub 2021 Jan 16. PMID 33602603

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 37 subjects were enrolled. 8 subjects failed screening. 16 were randomized to either the Biotene then placebo arm and 13 were randomized to the water then Biotene arm.
Groups:
- Biotene Then Placebo: People who present with dry mouth and will receive a single dose of Biotene.
  Biotene: Biotène Dry Mouth Moisturizing Spray contains water, polyglycitol, propylene glycol, sunflower oil, xylitol, milk protein extract, potassium sorbate, acesulfame K, potassium thiocyanate, lysozyme, lactoferrin, lactoperoxidase. 3 sprays, approximately 15 mL.
- Placebo Then Biotene: People who present with dry mouth and will receive a single dose of an alternative agent.
  Placebo: IND/IDE exempt device primarily water
Period: First Intervention
Arm/Group | Biotene Then Placebo | Placebo Then Biotene
Started | 16 | 13
Completed | 14 | 12
Not Completed | 2 | 1
Period: Washout
Arm/Group | Biotene Then Placebo | Placebo Then Biotene
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Biotene Then Placebo | Placebo Then Biotene
Started | 14 | 12
Completed | 14 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Biotene Then Placebo | Placebo Then Biotene | Total
Number analyzed (Participants) | 16 | 13 | 29
Age, Categorical [Count of Participants; unit: Participants] — Population: One participant did not have data collected for age in the Biotene then Placebo arm.
  Participants
    number analyzed (Participants) | 15 | 13 | 28
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 9 | 10 | 19
    >=65 years | 6 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 9 | 21
  Male | 4 | 4 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 15 | 13 | 28
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 2 | 6
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 16 | 13 | 29

OUTCOME MEASURES:

1. Primary Outcome: Mean Duration of Action of Intervention
Description: Participant will receive a dose of Biotene or placebo (water) and will be asked if their mouth is dry up to 2 hrs. The time at which their mouth becomes dry again will be the duration of action.
Time Frame: baseline up to 2 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Biotene | Placebo
Number analyzed (Participants) | 26 | 26
minutes | 27 (25) | 26 (25)

2. Secondary Outcome: Mean Tolerability of Product
Description: Subjects were asked to agree or disagree with the following statement where 1= strongly agree and 5- strongly disagree: The taste of the product was tolerable.
Time Frame: 2 hours
Population: Data from 1 subject was excluded due to inability to comprehend the instructions for rating xerostomia-related oral discomfort.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biotene | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | 4.2 (0.9) | 3.8 (1.3)

3. Secondary Outcome: Mean Acceptability of Product
Description: Subjects were asked to agree or disagree with the following statement where 1= strongly agree and 5- strongly disagree: The thickness of the product was acceptable.
Time Frame: 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biotene | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | 4.2 (0.9) | 3.9 (1.1)

4. Secondary Outcome: Mean Continued Use of Project
Description: Subjects were asked to agree or disagree with the following statement where 1= strongly agree and 5- strongly disagree: I would like to continue using this product.
Time Frame: 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biotene | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | 3.1 (1.1) | 2.9 (1.0)

5. Secondary Outcome: Mean Purchase Product Rating
Description: Subjects were asked to agree or disagree with the following statement where 1= strongly agree and 5- strongly disagree: I would purchase this product to use on a regular basis.
Time Frame: 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biotene | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | 2.9 (1.1) | 2.6 (0.9)

6. Secondary Outcome: Mean Ease of Use of Product
Description: Subjects were asked to agree or disagree with the following statement where 1= strongly agree and 5- strongly disagree: This product is easy to use.
Time Frame: 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biotene | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | 4.0 (0.8) | 3.9 (0.8)

7. Secondary Outcome: Mean Preference for Another Product
Description: Subjects were asked to agree or disagree with the following statement where 1= strongly agree and 5- strongly disagree: I would prefer using another product.
Time Frame: 2 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Biotene | Placebo
Number analyzed (Participants) | 25 | 25
score on a scale | 3.2 (0.9) | 3.4 (0.9)

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | Biotene | Placebo
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/29
Other Adverse Events (participants affected / at risk) | 0/29 | 0/29

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2019-07-05): https://cdn.clinicaltrials.gov/large-docs/31/NCT03663231/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2020-05-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT03663231/Prot_SAP_001.pdf